CLINICAL TRIAL: NCT02117622
Title: A Multi-centre, Prospective, Open-label, Single-arm, Non-interventional, Post Marketing Surveillance (PMS) Study of Tresiba® (Insulin Degludec) to Evaluate Long Term Safety and Efficacy in Patients With Diabetes Mellitus in Routine Clinical Practice in India
Brief Title: A Non-interventional, Post Marketing Surveillance (PMS) Study of Tresiba® (Insulin Degludec) to Evaluate Long Term Safety and Efficacy in Patients With Diabetes Mellitus in Routine Clinical Practice in India
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1250-4129; U1111-1145-9828 (Other: WHO); ENCEPP/SDPP/6318 (Registry Identifier: EU PASS)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with diabetes mellitus requiring insulin therapy
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Treatment according to routine clinical practice at the discretion of the treating physician. The assignment of the patient to Tresiba® is decided in advance of this study

SUMMARY:
This study is conducted in Asia. The aim of the study is to evaluate long term safety and efficacy of Tresiba® (insulin degludec) in patients with diabetes mellitus in routine clinical practice in India.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities (Study related activities are any procedure related to recording of data according to the protocol). The historical data including the data before informed consent obtained (e.g. glycosylated haemoglobin (HbA1c), fasting plasma glucose (FPG), severe hypoglycaemia before the start of Tresiba® therapy) can be used for baseline data
* Patients with insulin requiring diabetes mellitus and who is scheduled to start treatment with Tresiba® based on the clinical judgment of their treating physician

Exclusion Criteria:

* Known or suspected allergy to Tresiba®, the active substance or any of the excipients
* Previous participation in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Patients who are or have previously been on Tresiba® therapy
* Patients who are participating in other studies or clinical trials
* Patients who are pregnant, breast feeding or have the intention of becoming pregnant within the following 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus requiring insulin therapy who qualify for starting treatment with Tresiba® based on the clinical judgment by their treating physician during enrolment period.
Sampling Method: Non-Probability Sample
Enrollment: 1056 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) by preferred term | During 1 year of treatment

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAEs) by preferred term | During 1 year of treatment
Incidence of serious adverse drug reactions (SADRs) by preferred term | During 1 year of treatment
Incidence of adverse drug reactions (ADRs) by preferred term | During 1 year of treatment
Incidence of severe hypoglycaemia | During 1 year of treatment
Change from baseline in glycosylated haemoglobin (HbA1c) | Baseline (Visit 1, week 0), end of study (Visit 4, week 52)
Change from baseline in fasting plasma glucose (FPG) | Baseline (Visit 1, week 0), end of study (Visit 4, week 52)
Incidence of confirmed hypoglycaemia | During 1 year of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (24):
- India (24):
  - Novo Nordisk Investigational Site, Guntur, Andhra Pradesh
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Vijayawada, Andhra Pradesh
  - Novo Nordisk Investigational Site, Guwahati, Assam
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Ghuma, Gujarat
  - Novo Nordisk Investigational Site, Gurgaon, Haryana
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Thrissur, Kerala
  - Novo Nordisk Investigational Site, Bhopal, Madhya Pradesh
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Nagpur, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Delhi, New Delhi
  - Novo Nordisk Investigational Site, Mohali, Punjab
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Coimbatore, Tamil Nadu
  - Novo Nordisk Investigational Site, Madurai, Tamil Nadu
  - Novo Nordisk Investigational Site, Noida, Uttar Pradesh
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Chennai
  - Novo Nordisk Investigational Site, New Delhi
  - Novo Nordisk Investigational Site, Thriruvananthapuram

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com